CLINICAL TRIAL: NCT05911204
Title: Prevalence of Women Exposed to Intense and Prolonged Noises During the 3rd Trimester of Pregnancy
Brief Title: Exposure to Intense and Prolonged Noises During Pregnancy
Acronym: GestaNoise
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Michel HASCOET, Professor, Central Hospital, Nancy, France
Other Study IDs: 2023-A00588-37
Record Dates: First submitted 2023-06-09; First posted 2023-06-20 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Noise Exposure
Keywords: Pregnancy; Intense and prolonged noise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mothers: One single group of mothers exposed to intense and sustained noises during pregnancy
  Interventions: Other: Questionnaire about intense noises exposure during pregnancy

INTERVENTIONS:
Other: Questionnaire about intense noises exposure during pregnancy — Response to questionnaire given within 3 days after delivery about noise exposure

SUMMARY:
Hearing is an essential element for the development of language and conditions an appropriate cognitive, psychological and social development of children. Therefore, congenital deafness represents a real public health problem, justifying the implementation of a national neonatal screening for hearing disorders in newborns.

The intensity at which the fetus perceives sound at 27-29 weeks of amenorrhea (SA) is about 40 decibels (dB), it recognizes its mother's voice from the 33rd SA, and then its perception capacity evolves to the adult level at term. These data suggest that the fetus is sensitive to its sound environment from the 3rd trimester of pregnancy. The development of hearing could be damaged in case of prolonged exposure to intense noise. Studies have demonstrated an harmful effects of long and sustained exposure to noise on hearing in adults. In addition, a recent survey showed that 40% of the population of Ile-de-France felt that noise had a significant impact on their health . The effects of prolonged loud noise exposure on human fetal hearing are not fully understood and few studies have assessed the prevalence of women exposed to loud and lengthy noise in a population of postpartum women. This study aims evaluating the prevalence and the impacte of an exposure to Intense and Prolonged Noises during Pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Woman who gave birth at the Nancy Regional Maternity Hospital
* Woman having received complete information on the organization of the research and not having objected to her participation and the use of her data
* Woman affiliated to a social security scheme or beneficiary of such a scheme
* Woman understanding French and able to complete a self-questionnaire or having the possibility of being assisted for the filling

Exclusion Criteria:

* Woman for whom a diagnosis of malformation or genetic anomaly of the fetus was established in the antenatal period

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All mothers above 18 years old who have given birth and are cared for at the Nancy Regional University Maternity will be offered a questionnaire upon their arrival in their room in the mother-child sector
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Exposure to Intense and Prolonged Noises during Pregnancy | Collected at the routine newborn discharge examination, 72 or 96 hours after delivery, depending on the type of delivery
  A questionnaire will be given to the mother within 3 days after delivery

SECONDARY OUTCOMES:
Impact of noise exposure during pregnancy on health status, qualitative variable | Collected at the routine newborn discharge examination, 72 or 96 hours after delivery, depending on the type of delivery,
  A questionnaire given to the mother collecting her feelings on the impact of noise (no; some; heavy)
Newborn hearing screening, binary variable (presence of hearing impairment, absence of hearing impairment) | Collected at the routine newborn discharge examination, 72 or 96 hours after delivery, depending on the type of delivery
  Collection of the results of the routine hearing screening of the infants (presence of hearing impairment, absence of hearing impairment)
Women's knowledge of the risk of noise exposure during pregnancy on newborn hearing impairment, binary variable | Collected at the routine newborn discharge examination, 72 or 96 hours after delivery, depending on the type of delivery, where existing data on newborn hearing screening will be collected
  a questionnaire given to the mother after the birth (yes or no)

CONTACTS AND LOCATIONS:
Locations (1):
- Maternite Regionale Universitaire CHRU NANCY, Nancy, Lorraine, France